CLINICAL TRIAL: NCT05923853
Title: Electronic Optimization of Inspired Oxygen During Mechanical Ventilation, a Pragmatic Randomized Trial
Brief Title: Electronic Optimization of Inspired Oxygen During Mechanical Ventilation, a Pragmatic Randomized Trial (OPTI-Oxygen)
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: DSMB review pending
Sponsor: Ohio State University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Sonal Pannu, Associate Professor of Internal Medicine, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2023H0016
Record Dates: First submitted 2023-06-05; First posted 2023-06-28 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Hyperoxia
MeSH Terms: conditions — Hyperoxia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Respiratory therapists and study coordinators will be unblinded. Study investigators, medical monitor and statistician will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oxygen (FiO2) Titration per E-alerts (Experimental): All eligible mechanically ventilated patients, FiO2 titration and SpO2 goal range will be based on the correlation between SpO2 and arterial oxygen saturation (SaO2). E-alerts will be sent in the intervention arm as reminders for FiO2 titration.
  Interventions: Other: FiO2 titration using electronic alert system
- Oxygen Titration per Standard of Care (No Intervention): In the control arm, patients will have oxygen titrated per current standard of care (SpO2=88-92%, titrate FiO2 at least every 4 hours). Physician place oxygen titration orders in EMR and respiratory therapists conduct FiO2 titration without electronic alerts.

INTERVENTIONS:
Other: FiO2 titration using electronic alert system — In the intervention arm, arterial oxygen saturation (SaO2) and peripheral oxygen saturation (SpO2) will be initially noted. Based on the correlation between the SaO2 and SpO2 the optimal oxygenation range will be determined. E-alerts will then be used to monitor oxygenation for patients in the intervention arm, based on SpO2 values generated by the patient due to the FiO2 given to the patient through the ventilator. Once an e-alert is sent, the respiratory therapist has 45 minutes for adjusting oxygen. Then the e-alert continues to monitor FiO2 and SpO2 values in this manner for every 45 minute period until the ventilator is attached to the patient.
  Arms: Oxygen (FiO2) Titration per E-alerts

SUMMARY:
OPTI-Oxygen is a single center, stepped wedged, cluster-randomized, un-blinded, pragmatic, comparing the use of a combined inspired oxygen (FiO2) and peripheral oxygen saturation (SpO2) titration strategy utilizing electronic health records (EHR) based electronic alerts (e-alerts) for respiratory therapists in mechanically ventilated critically ill adults. All eligible mechanically ventilated patients, FiO2 titration and SpO2 goal range will be based on the correlation between SpO2 and arterial oxygen saturation (SaO2). E-alerts will be sent in the intervention arm as reminders for FiO2 titration. In the control arm, patients will have oxygen titrated per current standard of care (SpO2=88-92%, titrate FiO2 at least every 4 hours).

DETAILED DESCRIPTION:
We will conduct a single center, stepped wedged, cluster-randomized, un-blinded, pragmatic, comparing the use of a combined inspired oxygen (FiO2) and peripheral oxygen saturation (SpO2) titration strategy utilizing electronic health records (EHR) based electronic alerts (e-alerts) for respiratory therapists in mechanically ventilated critically ill adults. The participating intensive care units (ICU) will be medical, cancer, surgical (general surgery and trauma) and coronary critical care at the Ohio State University, Wexner Medical Center and James Cancer Hospital (128 beds). In this stepped wedge design, there will be nested randomization. A 12-13 bed pod within each of the 4 ICU's will be randomized as "step". Each 12-13 bed pod, geographically located within a unit will serve as a cluster and transition from control to intervention will occur every 6 weeks, with an initial 2 week implementation period. All intubated patients meeting inclusion criteria in a particular cluster will be in the intervention or control group per the assignment of that cluster. In the intervention arm, arterial oxygen saturation (SaO2) and peripheral oxygen saturation (SpO2) will be initially noted. Based on the correlation between the SaO2 and SpO2 the optimal oxygenation range will be determined. Then E-alerts will be used to monitor oxygenation for patients in the intervention arm, based SpO2 values generated by the patient due to the FiO2 given to the patient through the ventilator. E-Alerts search for SpO2 and FiO2 values every minute to evaluate if they meet criteria for optimal oxygenation. If in a 45 minute period 80% of values for both SpO2 and FiO2 values are do not meet target range then an e-alert (text message) is sent to the respiratory therapy cisco phones recommending that oxygen needs to be titrated. Once an e-alert is sent, the respiratory therapist has 45 minutes for adjusting oxygen. Then the e-alert continues to monitor FiO2 and SpO2 values in this manner for every 45 minute period until the ventilator is attached to the patient. (Details in study procedures, section 5). In the control arm, FiO2 titration will be assessed by the optimal oxygenation criteria by current standard of care. This is done by following the ICU ventilator management guidelines. Per the ventilator management guidelines assessment for FiO2 titration is recommended at least once in 4 hours to maintain oxygenation with the optimal range. Treatment allocation (SpO2 and FiO2 targeted titration) will cross over to a new cluster at the conclusion of each period. Protocol adherence will be monitored. Data will be collected until hospital discharge. The study will be carried about with waiver of consent, because the target ranges studied are used as part of routine clinical care in the ICU, and are interventions to which patients would be exposed even if not participating in the study. There is clinical equipoise, i.e. have inadequate prior data to suggest the superiority of one approach over the other. Additionally, patients in the trial would be expected to receive similar oxygen therapy in an unstructured manner if they were not in the trial.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Presence of mechanical ventilation

Exclusion Criteria:

* Pregnancy
* Prisoner status
* Pneumothorax
* Carbon monoxide poisoning
* Hyperbaric oxygen therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 936 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of time during mechanical ventilation spent within the target range, SpO2 of 90-94% (conservative) or SpO2 of 93-97% (liberal) at any FiO2 in respective algorithms. | through study completion, average of 28-30 days
  Percent time during mechanical ventilation in target range.

SECONDARY OUTCOMES:
Proportion of time with SpO2 > 94% or SpO2 > 97% with FiO2 ≤ 0.4 in respective algorithms. | through study completion, average of 28-30 days
  Percent time during mechanical ventilation above target range.
Proportion of time with time with SpO2 < 90% or SpO2 < 93% in respective algorithms. | through study completion, average of 28-30 days
  Percent time during mechanical ventilation below target range.
Length of ICU stay | through study completion, average of 28-30 days
  Total number of days in the ICU.
Length of hospital stay | through study completion, average of 28-30 days
  Total number of days in the hospital.
Hospital mortality | through study completion, average of 28-30 days
  Dead or alive at hospital discharge.
Ventilator-Free Days | through study completion, average of 28-30 days
  Alive and free from ventilator support at day 28.
Vasopressor-Free Days | through study completion, average of 28-30 days
  Alive and free from vasopressor support at day 28.
ICU-Free Days | through study completion, average of 28-30 days
  Alive and out of the ICU at day 28.
New onset arrhythmia when SpO2<90% | through study completion, average of 28-30 days
  Arrhythmia onset during hypoxemia.
Change to comfort care status (DNRCC) and time to DNRCC after enrollment. | until hospital discharge or death befoe hospital discharge, upto 60 days
  Change to comfort care status after enrollment will be recorded and analyzed as a dichotomous outcome. Time to DNRCC after enrollment will be evaluated in an exploratory nature using appropriate time-to-event models. Hospital mortality while in comfort care status will also be examined as an exploratory endpoint.

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified dataset will be shared after the completion of data analysis of the last patient is enrolled.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 1 year after enrollment of the last patient. Data will be available for 5 years
Access Criteria: To be determined

REFERENCES:
- [Derived] Pannu SR, Peters J, Zimmer J, Brock GN, Exline M, Horowitz JC, Thompson TB, Rice TW, Crouser ED. Optimization of Inspired Oxygen during Mechanical Ventilation (OPTI-OXYGEN): rationale and design of a pragmatic randomised controlled trial. BMJ Open. 2025 Jun 5;15(6):e094924. doi: 10.1136/bmjopen-2024-094924. PMID 40473278